CLINICAL TRIAL: NCT01516021
Title: Fat Intake Modulates Cerebral Blood Flow in Homeostatic and Gustatory Brain Areas in Humans
Brief Title: How Fat Influences the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other); German Federation of Industrial Research Associations (Other); Zentrum für Ernährungsmedizin und Prävention (Other); German Center for Diabetes Research (Other); University of Hohenheim (Other)
Responsible Party: Principal Investigator, Sabine Frank, Principal Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: YOG
Record Dates: First submitted 2012-01-09; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Fat Processing in the Brain
Keywords: Fat ingestion; hypothalamus; insula; fMRI; CBF

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- high fat yoghurt intake (Experimental): 500 ml of a high fat yoghurt
  Interventions: Dietary Supplement: intake of high or low fat yoghurt
- low fat yoghurt intake (Experimental)
  Interventions: Dietary Supplement: intake of high or low fat yoghurt

INTERVENTIONS:
Dietary Supplement: intake of high or low fat yoghurt — intake of 500 ml of a high fat yoghurt on one day and intake of 500 ml of a low fat yoghurt on the other day

SUMMARY:
The aim of the current study was to investigate the effect of a high versus a low fat meal (operationalized by high and low fat yoghurt) on homeostatic and gustatory brain regions.

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy

Exclusion Criteria:

* lactose intolerance
* fMRI contraindications (metal implants,...)

Ages: 25 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Changes in Cerebral Blood Flow due to the high or low fat yoghurt intake after 30 minutes and 120 minutes compared to a baseline measurement 30 minutes before yoghurt intake. | 30 minutes before as well as 30 minutes and 120 minutes after fat intake
  We were interested in differential brain activations due to the high or low fat meal. To assess this, the mentioned time points are suitable.
  The Cerebral Blood Flow is measured using Arterial Spin Labeling sequences in a functional magnetic resonance tomography.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Tuebingen, MEG Center, Tübingen, Germany

REFERENCES:
- [Derived] Frank S, Linder K, Kullmann S, Heni M, Ketterer C, Cavusoglu M, Krzeminski A, Fritsche A, Haring HU, Preissl H, Hinrichs J, Veit R. Fat intake modulates cerebral blood flow in homeostatic and gustatory brain areas in humans. Am J Clin Nutr. 2012 Jun;95(6):1342-9. doi: 10.3945/ajcn.111.031492. Epub 2012 May 9. PMID 22572644